CLINICAL TRIAL: NCT01050478
Title: Open-label, Single Arm, Interventional Study to Explore the Efficacy and Safety of Paliperidone ER in the Management of Patients With Acute Agitation and/or Aggression
Brief Title: IMPACT: A Study to Explore the Efficacy and Safety of Paliperidone ER in Patients With Acute Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015427; R076477SCH3038 (Other: Janssen); 2009-015629-35 (EudraCT Number)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Psychomotor Agitation; Acute Disease
Keywords: acute agitation; aggression; psychosis; paliperidone extended release
MeSH Terms: conditions — Psychomotor Agitation; Acute Disease; Aggression; Psychotic Disorders | interventions — Paliperidone Palmitate; Benzodiazepines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone ER (Experimental): Paliperidone ER: recommended dose: 6 mg/day. Can be 9 mg/day for patients with an acute exacerbation of schizophrenia. A benzodiazepine for sedation and/or rescue medication can be added with a maximum of 7.5 mg/day, at the investigators' discretion.
  Interventions: Drug: Paliperidone ER; Drug: Benzodiazepine

INTERVENTIONS:
Drug: Paliperidone ER — paliperidone ER at 2 dosage levels (6 and 9 mg/day)
Drug: Benzodiazepine — Participants may receive the benzodiazepine lorazepam [0-7.5 milligram (mg) per day] as needed for sedation or rescue medication at the investigator's discretion.

SUMMARY:
This study will investigate the effect of paliperidone ER (in combination with or without benzodiazepines) in patients presenting with symptoms of agitation and/or aggression in the context of psychosis, and will generate data regarding both efficacy and safety in the acute setting.

DETAILED DESCRIPTION:
Psychomotor agitation that requires hospitalization is a common event during the course of certain major psychiatric disorders, including schizophrenia. Emergency psychiatric services are the first doorway for the control of agitation and behavioural disturbances of the mentally ill in order to avoid dangerousness and aggression towards themselves and/or others. The use of drugs that influence the psychological behaviour (psychotropic drugs) should help to handle agitation and aggression, rapidly rendering people calm and/or sedated without producing distressing or dangerous adverse events, and facilitating extended assessment and definitive treatment. Oral atypical antipsychotics, alone or in combination with a benzodiazepine, are considered first line treatment for patients who present at the emergency ward with mild to moderate psychotic agitation. Paliperidone is a new atypical antipsychotic therapeutic agent for the treatment of schizophrenia. Paliperidone extended release (ER) might be considered as a treatment option for patients presenting with agitation and/or aggression (in combination with short term use of benzodiazepines) because of its fast onset of action and limited or no long term sedating effects. This open-label, single arm, multicenter, interventional descriptive study will collect data on efficacy and safety during first days of treatment with paliperidone ER in patients with acute agitation in the context of psychosis in the psychiatric emergency setting. The assessment of effectiveness/response will be based on Positive And Negative Syndrome Score Exciting Component (PANSS-EC) improvement. Safety evaluations include the incidence of serious and non-serious adverse events. The study will end after 5 days of treatment or at day of discharge from the hospital, whatever comes first. 6 mg (patients with an acute exacerbation of schizophrenia in a real-world setting an initial dose of paliperidone 9 mg once daily may provide optimal clinical efficacy with good tolerability) tablet, oral, once a day during the study duration (5 days).

ELIGIBILITY:
Inclusion Criteria:

Patient presenting with acute agitation and/or aggression in the context of psychosis, suspected schizophrenia PANSS-EC score >=20 Patient is outpatient in need of hospitalization female patients of childbearing potential must have a negative urine pregnancy test at baseline and further adequate anticonceptive protection signed informed consent

Exclusion Criteria:

Received benzodiazepines 4 hours prior to enrolment Received antipsychotic medication 72 hours prior to enrolment agitation, aggression or violent behaviour that necessitates the use of intramuscular or intravenous medication Patient's preference for intramuscular or intravenous medication Patient judged to be at high risk for suicidal behaviour Pregnant or breast feeding females Patient received clozapine or long-acting injectable antipsychotic during the last 3 months Serious unstable medical condition, including known clinically relevant lab abnormalities History of current symptoms or tardive dyskinesia History of neuroleptic malignant syndrome Participation in an investigational drug trial in the 30 days prior to selection Inability to swallow the study medication whole with the aid of water (chewing, dissolving, dividing or crushing the study medication is not allowed) Patients with a narrowing or blockage of their gastro-intestinal tract Patients with current or known history (past 6 months) of substance dependence according to DSM-IV criteria known hypersensitivity to paliperidone ER or risperidone Employees of the investigator or study centre, persons with direct involvement in the proposed study or other studies under the direction of that investigator or study centre, or family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients having an improvement of 40% or more on PANSS-EC | All of the 8 study visits during the 5-day study duration

SECONDARY OUTCOMES:
Assessing the change from baseline on PANSS-EC (Positive and Negative Syndrome Scale - Exciting Component) | All of the 8 study visits during the 5-day study duration
Assessing the change from baseline on the OAS (Overt Agression Scale) | All of the 8 study visits during the 5-day study duration
Assessing disease severity (Global Assessment of Functioning) | All of the study visits during the 5-day study duration, except study visit 2
Assessing daytime drowsiness (Behaviour Activity Rating Scale) | All of the 8 study visits during the 5-day study duration
Assessing tolerability and safety by reporting adverse events and vital signs | All of the 8 study visits during the 5-day study duration

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.
Locations (14):
- Belgium (14):
  - Bruges
  - Brussels
  - Dave
  - Diest
  - Ghent
  - Henri-Chapelle
  - Heusden
  - Kortrijk
  - La Louvière
  - Liège
  - Marchienne-au-Pont
  - Ottignies
  - Sint-Denijs-Westrem
  - Tournai

REFERENCES:
- [Result] Audenaert K, Godenir F, Geerts P, Van Gils L, Wouters C, Detraux J. IMPACT (Invega in the Management of Patients in the ACute seTting): results from a Belgian study using paliperidone extended-release in the management of psychotic patients with acute agitation and/or aggression. Acta Psychiatrica Belgica 2013 113 (4) 21-30.
- See also: Open-label, single arm, interventional study to explore the efficacy and safety of paliperidone ER in the management of patients with acute agitation and/or aggression — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=250&filename=CR015427_CSR.pdf